CLINICAL TRIAL: NCT06363526
Title: Effectiveness of 5-week Digital Respiratory Practice in a Group of Children With Duchenne Muscular Dystrophy and Becker Muscular Dystrophy.
Brief Title: Effectiveness of 5-week Digital Respiratory Practice in Children With Duchenne and Becker Muscular Dystrophies.
Acronym: DMDrespy2024
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Rocío Martín Valero, Principal Investigator, University of Malaga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMalagaDRIP
Record Dates: First submitted 2024-03-22; First posted 2024-04-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Breathing exercises; Inspiratory muscle training; Pulmonary rehabilitation; Expiratory muscle training
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Intervention Model Description: 12 participants were randomized to follow a digital respiratory physiotherapy program for 5 weeks. The participants were evaluated at the beginning and at the end of the study, and the results will be measured before and after each intervention during the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Duchenne muscular dystrophy and Becker muscular dystrophy (Experimental): A group of 12 patients with Duchenne muscular dystrophy and Becker muscular dystrophy that will be following a digital respiratory physiotherapy program.
  Interventions: Other: Digital respiratory intervention program

INTERVENTIONS:
Other: Digital respiratory intervention program — A 4 times a week for a period of 5 weeks will be done, for a duration of 55-60 minutes (20 sessions), with an intensity adapted to the characteristics of each participant. Moreover, an intervention program will be used based on respiratory muscle training exercises, upper limb strength work, yoga, diaphragmatic awareness exercises, always trying to do them through the use of games, and even try to include exercises that use motor imagery.
  The intervention program is carried out and stimulated through videos and therapeutic teaching to the caregivers in the first evaluation session, as well as as well as with a weekly follow-up using WhatsApp or Zoom as forms of communication, or a telephone call to ensure correct follow-up of the intervention program. Moreover, YouTube videos, own videos prepared by the physiotherapy will be used to help optimally resolve doubts that arise when carrying out the program by video call.

SUMMARY:
The purpose of this study is to analyze the effectiveness of a 5-weeks respiratory digital intervention program in patients with Duchenne muscular dystrophy and Becker muscular dystrophy.

DETAILED DESCRIPTION:
It will be done 4 times a week for a period of 5 weeks, for a duration of 55-60 minutes (20 sessions), with an intensity adapted to the characteristics of each participant. An intervention program will be used based on respiratory muscle training exercises, upper limb strength work, yoga, diaphragmatic awareness exercises, always trying to do them through the use of games, and even try to include exercises that use motor imagery.

It is advisable during intervention program to have a playful environment stimulated for the children, and that the intervention program is carried out and stimulated through videos and therapeutic teaching to the caregivers in the first evaluation session, as well as with a weekly follow-up using WhatsApp as forms of communication, or a telephone call to ensure correct follow-up of the intervention program.

It is essential that to carry out the intervention, videos obtained from YouTube, own videos prepared to explain the exercises in a playful way applied to children, and even other applications such as Spotify to work with music, will be used, being offered in case of Zoom calls may be necessary to help optimally resolve doubts that arise when carrying out the program by video call.

At the end of the respiratory digital physiotherapy program, variables will be evaluated by the principal examiner.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Duchenne muscular dystrophy and patients with Becker muscular dystrophy will be chosen.
* Aged between 5 and 20 years.
* Child who could walk and follow the intervention program, and were diagnosed according to the International Classification of Diseases, 10 Revision. code (G71-01); and who had an NSSA score greater than 20.

Exclusion Criteria:

* Patients who present associated heart disease.
* Patients who presentor fractures, a heart rate greater than 120 beats per minute, or an oxygen saturation less than 89% will be excluded.
* Participants who do not have the capacity to have internet at home to perform the intervention, as well as all patients whose caregivers did not agree to sign the informed consent.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Analyze the improvement of the forced vital capacity (FVC). | Baseline, up to 5 weeks.
  Forced vital capacity is a respiratory parameter which is obtained from spirometry and which provides objective, valid information. It will be performed using spirometry before and after the digital respiratory intervention program. The spirometer that will be used is the "EasyOne Air Spirometer that complies with ISO 26782 standards, following the national spirometric recommendations of the ATS/ERS 2019.

SECONDARY OUTCOMES:
Perform an anthropometric study of the patient's characteristics, taking into account weight; and also a general physical examination. | Baseline, up to 5 weeks.
  An anthropometric study of the patient's characteristics will be carried out, taking into account age, weight, as well as the average values that should be established based on age; as well as a general physical examination of the patient to analyze if they will be considered fit or not to carry out the program.
  The weight will be check by "SECA 700 MECHANICAL COLUMN SCALE WITH SECA 220 STADIOMETER", and the height will be analyze by a measuring tape.
Perform an anthropometric study of the patient's characteristics, taking into account age. | Baseline, up to 5 weeks.
  An anthropometric study of the patient's characteristics will be carried out, taking into account age, as well as the average values that should be established based on age; as well as a general physical examination of the patient to analyze if they will be considered fit or not to carry out the program.
Perform an anthropometric study of the patient's characteristics, taking into account height. | Baseline, up to 5 weeks.
  An anthropometric study of the patient's characteristics will be carried out, taking into account height, as well as the average values that should be established based on age; as well as a general physical examination of the patient to analyze if they will be considered fit or not to carry out the program.
Perform an anthropometric study of the patient's characteristics, taking into account sex. | Baseline, up to 5 weeks.
  An anthropometric study of the patient's characteristics will be carried out, taking into account height, as well as the average values that should be established based on sex; as well as a general physical examination of the patient to analyze if they will be considered fit or not to carry out the program.
Examine changes in forced expiratory pressure | Baseline, up to 5 weeks.
  Forced expiratory pressure is a respiratory parameter obtained through spirometry, which provides important information about the patient's respiratory status. Measuring it will be done with the same characteristics as that previously mentioned in the FVC.
Analyze changes in maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP). | Baseline, up to 5 weeks.
  Changes in the strength of the inspiratory and expiratory muscles will be assessed using a pressure meter with a reading range of ±300 cm H20 and an accuracy of 3% (MicroRPM® model, Vyaire Medical GmbH, Hoechberg, Germany) following the national recommendations of the Spanish Society of Pulmonology and Thoracic Surgery (SEPAR) (16).
Check if there are changes in the sniff nasal inspiratory pressure (SNIP) | Baseline, up to 5 weeks.
  The existence of changes in the diaphragm force index is assessed, measuring it in exactly the same way as the MIP and PEM.
Evaluate the fatigue in patients using an EPInfant test. | Baseline, up to 5 weeks.
  The amount of effort the child perceives during the sessions is assessed. It shows 11 descriptors numbered from 0 to 10 and 5 verbal descriptors located every 2 levels of the numbered descriptors, along with a drawing of a child doing physical activity in an increasing manner, increasing in intensity from left to right. The higher the numerical value, the worse the result is considered.
Evaluate the quality of life of patients using a scale called "Kindscreen-52". | Baseline, up to 5 weeks.
  52-item scale carried out in Ravens-Sieberer U and validated in Spanish by Rajmil L, which assesses physical and psychological well-being, mood and emotions, self-perception, autonomy and relationship with friends and social life. . The scores were transformed into a scale from 0 to 100 to facilitate their interpretation: the higher the score, the higher HRQoL.
North Star Ambulatory Assessment o NSAA | Baseline, up to 5 weeks.
  Designed to capture the construct of ambulatory function in DMD. 17-item scale that grades performance of various functional skills on a scale from 0 (unable), 1 (completes independently but with modifications), and 2 (completed without compensation). Total score 0 - 34 with a higher score denoting a higher level of function. It includes two timed tests. Timed rise from floor (RFF) and timed 10 metre walk / run test (10MWR). Validated and regularly used in clinical trials as well as clinic. Well understood by families. The best score is 34 points.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Martín-Valero, PhD, Study Director — University of Malaga
Locations (1):
- Rocío Martín-Valero, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No